**Study Title:** Umbilical Trocar Site Is the Usual Suspect for Trocar Hernia After Laparoscopic

Cholecystectomy: A Prospective Study

**NCT ID:** Not yet assigned.

**Date:** April 15, 2025

# **CLINICAL STUDY REPORT (CSR)**

Study Title: Umbilical Trocar Site Is the Usual Suspect for Trocar Hernia After Laparoscopic

Cholecystectomy: A Prospective Study

Study Type: Prospective, randomized controlled trial

**Study Duration:** April 15, 2022 – June 15, 2024

Study Location: Umraniye Training and Research Hospital, Department of General Surgery

Principal Investigator: Ass. Prof. Dr. Tolga Canbak

ClinicalTrials.gov ID: Not yet assigned

### 1. Study Synopsis

## **Objective:**

To evaluate whether the site of gallbladder retrieval (umbilical vs. epigastric) affects the incidence of trocar site hernia (TSH) following laparoscopic cholecystectomy (LC), and to identify risk factors for TSH.

### Design:

Prospective, randomized, single-blind, controlled study with two parallel arms.

### **Participants:**

110 patients undergoing elective LC for gallstone disease were randomized. After accounting for conversions and loss to follow-up, 100 patients (50 in each group) were included in the final analysis.

#### **Intervention:**

Standard 4-port LC performed. Gallbladder retrieved via either:

Group U: Umbilical trocar (10 mm)

Group E: Epigastric trocar (10 mm)

**Primary Outcome:** 

Incidence of trocar site hernia at 12-month follow-up.

## **Secondary Outcomes:**

Gallbladder retrieval time

Postoperative pain scores (VAS at 6 and 24 hours)

Risk factor analysis for TSH development

# **Key Results:**

TSH occurred in 12% (6/50) of umbilical group and 10% (5/50) of epigastric group (P = 1.00).

All hernias were located at the umbilical site.

Epigastric retrieval was faster (P = 0.013) but associated with more early pain (P = 0.027).

Fascial widening was the only independent risk factor for TSH (OR = 4.08, P = 0.05).

## 2. Study Design

#### Randomization:

Performed via the Alea Randomisation mobile app. Allocation was sealed and revealed intraoperatively before specimen retrieval.

### **Blinding:**

Patients were blinded. Surgeons were not blinded due to the nature of the procedure, but were unaware of group allocation until extraction.

### **Surgeon Consistency:**

All surgeries were performed by three experienced general surgeons using standardized techniques.

## **Antibiotic Prophylaxis:**

Intravenous cefazolin 2 g administered preoperatively.

#### 3. Inclusion / Exclusion Criteria

### **Inclusion:**

 $Age \ge 18$ 

Gallstone disease

No significant systemic comorbidities

#### **Exclusion:**

Age < 18

Conversion to open surgery

Acute cholecystitis

Prior common bile duct surgery

Presence of diastasis recti or umbilical hernia

## 4. Surgical Technique

Standard LC using:

10 mm umbilical camera port

10 mm epigastric port

Two 5 mm subcostal ports

Fascial closure was performed only at the umbilical site using polyglactin sutures.

Epigastric port sites were not sutured.

Gallbladder retrieval performed using a bag.

## 5. Postoperative Management & Follow-Up

### **Pain Control:**

IV paracetamol and tramadol postoperatively. VAS recorded at 6 and 24 hours.

## Discharge & Follow-up:

Routine discharge on Day 1 if no complications. All patients followed for 12 months.

## Hernia Diagnosis:

Symptomatic patients evaluated with ultrasonography. Asymptomatic patients underwent scheduled USG at 6 and 12 months.

### 6. Statistical Analysis

- Data analyzed with SPSS v26 and RStudio.
- Categorical data were analyzed using Fisher's exact or Chi-square tests
- Continuous variables were compared using Student's t-test or Mann–Whitney U test
- Univariate and multivariate logistic regression performed to evaluate TSH risk factors.
- Significance threshold: P < 0.05

## 7. Results Summary

### **Demographics:**

Age, BMI, and other baseline factors were comparable between groups.

#### **Outcomes:**

- Hernia rate: 6 in Group U, 5 in Group E (all at umbilicus)
- Retrieval time shorter in Group E (P = 0.013)
- Pain lower in Group U at 6h (P = 0.027)
- No difference in 24h VAS scores
- Multivariate Analysis:
- Fascial widening was the only independent predictor of TSH (OR = 4.08, P = 0.05)

#### 8. Discussion

- All trocar site hernias (TSH) occurred at the umbilical site, regardless of extraction route.
- This confirms the umbilicus as the most vulnerable location for hernia development after
- laparoscopic cholecystectomy.
- Epigastric extraction avoided direct stress on the umbilical site and was associated with no
- hernias at the epigastric port.
- Gallbladder retrieval was faster via the epigastric route, offering operative efficiency.
- Early postoperative pain (6h) was slightly higher with epigastric extraction but not clinically
- limiting.
- Fascial widening during extraction was the only independent risk factor for TSH.
- These findings support preferential use of the epigastric port for specimen retrieval to
- minimize hernia risk.

#### 9. Conclusion

While trocar site selection did not statistically alter the incidence of hernia, all hernias occurred at the umbilicus, highlighting its vulnerability. Fascial widening during extraction was a key modifiable risk factor. Epigastric retrieval may offer operative efficiency, but at a slight cost in postoperative discomfort.

## 10. Ethical Considerations

- Approved by the Clinical Research Ethics Committee of Istanbul University of Health
- Sciences, Umraniye Training and Research Hospital.
- All participants provided written informed consent.
- Study conducted in accordance with the Declaration of Helsinki.
- No funding received. No conflicts of interest declared.

# STATISTICAL ANALYSIS PLAN (SAP)

Study Title: Umbilical Trocar Site Is the Usual Suspect for Trocar Site Hernia After

Laparoscopic Cholecystectomy: A Prospective Study

Version: 1.0

**Prepared by:** Olgun ERDEM

Study Sponsor: Umraniye Research and Training Hospital

Principal Investigator: Ass. Prof. Dr. Tolga Canbak

## 1. Study Overview

This is a prospective, randomized, controlled clinical trial evaluating the incidence of trocar site hernia (TSH) in patients undergoing laparoscopic cholecystectomy, comparing gallbladder extraction via the umbilical versus epigastric port.

# 2. Study Objectives

# **Primary Objective:**

To assess whether the site of gallbladder retrieval (umbilical vs. epigastric trocar) affects the incidence of trocar site hernia.

### **Secondary Objectives:**

To compare postoperative pain levels at 6 and 24 hours between groups

To assess gallbladder retrieval time

To identify independent risk factors for the development of trocar site hernia

#### 3. Endpoints

## **Primary Endpoint:**

Incidence of trocar site hernia (clinical or ultrasonographic diagnosis within 12 months)

## **Secondary Endpoints:**

- Gallbladder retrieval time (in seconds)
- Visual Analogue Scale (VAS) pain scores at 6 and 24 hours postoperatively
- Occurrence of fascial widening and its association with TSH

Logistic regression model identifying independent risk factors for TSH

### 4. Analysis Populations

### **Intention-to-Treat (ITT):**

All randomized patients, excluding those who converted to open surgery or were lost to followup.

### Per Protocol (PP):

Patients who completed surgery and 12-month follow-up without major protocol deviations.

#### 5. General Statistical Methods

- Statistical significance threshold set at P < 0.05 (two-sided).
- All statistical analyses will be performed using SPSS v26.0 and RStudio v4.2.0.
- Results will be reported with appropriate confidence intervals (CIs) and effect sizes when
- applicable.

# 6. Data Handling and Assumptions

## **Missing Data:**

No imputation will be performed.

Patients lost to follow-up will be excluded from analysis of outcomes they did not complete.

#### **Outliers:**

Checked visually (boxplots, scatterplots).

No exclusions unless clinically justified.

## **Normality Testing:**

Shapiro-Wilk test used for continuous variables.

## 7. Baseline and Demographic Comparisons

Descriptive statistics: mean  $\pm$  SD for normally distributed data; median (min–max) for non-normal data; frequency (%) for categorical variables.

### **Comparisons:**

• Categorical variables: Chi-square or Fisher's exact test

• Continuous variables: Student's t-test or Mann–Whitney U test depending on distribution

# 8. Primary Endpoint Analysis

#### **Incidence of TSH:**

Compared between the umbilical and epigastric groups using Fisher's exact test.

## 9. Secondary Endpoint Analyses

- Gallbladder retrieval time: Compared using Mann–Whitney U test (non-normal distribution
- anticipated).
- Postoperative pain scores (VAS at 6h and 24h): Assessed separately at both time points.
- Compared using Mann–Whitney U test.
- Exploratory regression analyses: Univariate logistic regression to identify factors associated
- with TSH Variables with P < 0.2 or known clinical relevance will be entered into a
- multivariate logistic regression model.
- Odds Ratios (OR), 95% CI, and P-values will be reported.

### 10. Subgroup Analyses

Subgroup analysis will be performed for patients in the umbilical extraction group to evaluate the impact of fascial widening on TSH incidence using logistic regression.

### 11. Software

All analyses will be conducted using:

- SPSS v26.0 (IBM Corp., Armonk, NY, USA)
- RStudio v4.2.0 (The R Foundation)